# STUDY PROTOCOL

# TITLE: Process evaluation of the effectiveness of two transdiagnostic interventions targeting emotional regulation: compassion focused program and emotional skills training program

| N°ID RCB | N°CPP | N°CNIL |
|----------------|-----------------------------------|---------|
| 2020-A00551-38 | 2020.09.03 ter_<br>20.05.13.42837 | 2217007 |

Document date: 17/01/2021

| Promotor and investigator | Mathias BUTAUD, Psychiatrist 4 avenue Jean Perrot, 38000 Grenoble mathias_butaud@hotmail.com |
|---|---|
| Co-investigator | Céline BAEYENS Professor, Laboratoire Interuniversitaire de Psychologie (LIP/PC2S) Université Grenoble Alpes, UFR SHS, 1251 avenue Centrale, CS 40700, 38058 Grenoble Cedex 9 celine.baeyens@univ-grenoble-alpes.fr |
| Associated investigators | Rebecca BEGUE SHANKLAND Professor, Laboratoire Développement, Individu, Processus, Handicap, Education (DIPHE) Université Lyon 2, Bâtiment V (V211 à V216), 5, Avenue Pierre Mendès-France, 69676 Bron Cedex Rebecca.shankland@univ-grenoble-alpes.fr |
| | Marine PAUCSIK PhD Student and psychologist, laboratoire Interuniversitaire de Psychologie (LIP/PC2S) Grenoble Alpes, UFR SHS, 1251 avenue Centrale, CS 40700, 38058 Grenoble Cedex 9 Marine.paucsik@univ-grenoble-alpes.fr |
| | Dr Francis Gheysen Psychiatrist – Cabinet de psychiatrie 1, avenue du 6 juin, 14000 Caen fgheysen@aol.com |
| | Claire Cécile Périer Neuropsychologist – Centre Référent de Réhabilitation Psychosociale et de Remédiation cognitive (C3R) de Grenoble. Centre Ambulatoire de Santé Mentale, 8 place du Conseil de la Résistance, 38100 Saint-Martin-d'Hères ccperier@ch-alpes-isere.fr |

| | Rocio Roure Neuropsychologist – Centre Référent de Réhabilitation Psychosociale et de Remédiation cognitive (C3R) de Grenoble. Centre Ambulatoire de Santé Mentale, 8 place du Conseil de la Résistance, 38100 Saint-Martin-d'Hères rroure@ch-alpes-isere.fr |
|---|---|
| | Cécile Fluttaz Neuropsychologist – Centre Référent de Réhabilitation Psychosociale et de Remédiation cognitive (C3R) de Grenoble. Centre Ambulatoire de Santé Mentale, 8 place du Conseil de la Résistance, 38100 Saint-Martin-d'Hères cfluttaz@ch-alpes-isere.fr |
| | Sandrine Rebelle Neuropsychologist, Centre départemental de réhabilitation psychosociale des Glières 219 Chemin des bois des Fornets 74800 La Roche-sur-Foron 04 50 03 73 28 |
| Associated center | Centre Référent de Réhabilitation Psychosociale et de Remédiation cognitive (C3R) de Grenoble. Dr Benjamin Gouache Psychiatrist Centre Ambulatoire de Santé Mentale, 8 place du Conseil de la Résistance, 38100 Saint-Martin-d'Hères Bgouache@ch-alpes-isere.fr Centre départemental de réhabilitation psychosociale des Glières 219 |
| | Dr Céline Roussel Psychiatrist Chemin des bois des Fornets 74800 La Roche-sur-Foron 04 50 03 73 28 |
| Mandatary | Marine PAUCSIK PhD Student and psychologist - laboratoire Interuniversitaire de Psychologie (LIP/PC2S) Grenoble Alpes, UFR SHS, 1251 avenue Centrale, CS 40700, 38058 Grenoble Cedex 9 Marine.paucsik@univ-grenoble-alpes.fr |
| Scientific<br>Coordinators of the<br>Study - Clinical<br>Research Vigilance | Céline BAEYENS Professor, Laboratoire Interuniversitaire de Psychologie (LIP/PC2S) Université Grenoble Alpes, UFR SHS, 1251 avenue Centrale, CS 40700, 38058, Grenoble Cedex 9 celine.baeyens@univ-grenoble-alpes.fr |
| | Rebecca BEGUE SHANKLAND Professor, Laboratoire Développement, Individu, Processus, Handicap, Education (DIPHE) Université Lyon 2, Bâtiment V (V211 à V216), 5, Avenue Pierre Mendès- France, 69676 Bron Cedex Rebecca.shankland@univ-grenoble-alpes.fr |

#### Objectives:

The purpose of this research is to evaluate the effectiveness of two programs - Compassion Focused Program and Emotional Skills Training - on participants' emotional regulation, well-being, compassion, emotional skills, and anxiety-depressive symptoms compared to the control group in a subclinical population and clinical population

#### Types of studies:

- Multiple single-case study
- Randomized controlled study in subclinical population
- Pilot study in a clinical population

#### Primary Objectives:

Evaluation of the effectiveness of the Compassion Focused Program and Emotional Skills Training programs on participants' emotional regulation (DERS, Gratz & Roemer, 2004) compared to the control group.

#### Secondary objectives and criteria:

The secondary objectives are, in comparison to the control group, to evaluate (1) the effectiveness of the interventions on emotional regulation strategies (DERS, Dan-Glauser & Scherer, 2013), well-being (BE, Ryff, 1995, anxiety and stress symptoms (DASS21, Henry & Crawford, 2005), emotional competencies (S-PEC; Mikolajczak, Brasseur, & Fantini-Hauwel, 2014), and compassion (SCS; Neff, 2003) and (2) to assess program effectiveness processes on: feeling of effectiveness of emotional regulation (Bandura, 2006) and cognitive flexibility (CFI; Dennis & Vander Wal, 2010).

#### Control variables:

In addition to the primary and secondary objectives, we will control for two variables: participants' expectations of the intervention prior to the start of the program (QCA, Coste et al., 2019), and participants' satisfaction with the intervention at the end of the intervention (STTS-R, Oei & green, 2008).

#### Inclusion criteria

- Age between 18 and 65 years inclusive
- Person who can understand, speak and read French
- Person who was orally informed and gave informed consent to participate in the study
- Subject's participation in the study noted in the medical record

#### Non-inclusion criteria

- Participation in positive psychology, mindfulness or stress management groups for less than 3 months

- Change in psychotropic medication (taking, stopping, or changing dosage) within 2 months prior to study participation
- Person with a mental disability
- Person deprived of liberty by court order

### Numbers of subjects to be included:

- Single case study: 10 participants, 5 participants per group
- Randomized controlled study: 123 participants: 41 participants per group
- Pilot study: 60 patients, 20 patients per group

#### Provisional research schedule

| SINGLE CASE STUDY | |
|---|---|
| Beginning of inclusions | November 2020 |
| Inclusion period | 1 months |
| Duration of interventions | 3 months |
| Duration of participation for each subject | 5 months |
| Exclusion period (=period during which the participant will not be | |
| able to participate in any other research involving an emotional | 5 months |
| regulation intervention) | |
| RANDOMIZED CONTROLLED STUDY | |
| Beginning of inclusions | Février 2021 |
| Inclusion period | 18 mois |
| Duration of interventions | 3 mois |
| Duration of participation for each subject | 7 mois |
| Exclusion period (=period during which the participant will not be | |
| able to participate in any other research involving an emotional | 6 mois |
| egulation intervention) | |
| PILOT STUDY | |
| Beginning of inclusions | August 2021 |
| Inclusion period | 2 months |
| Duration of interventions | 3 mois |
| Duration of participation for each subject | 7 months |
| Exclusion period (=period during which the participant will not be | |
| able to participate in any other research involving an emotional | 6 months |
| regulation intervention) | |
| TOTAL RESEARCH TIME | 31 months |
| END OF THE RESEARCH | March 2022 |

#### Benefits for participants

The two interventions will allow individuals to become familiar with their emotions, to cope more easily with the emotional difficulties encountered in their daily lives and to develop new strategies to manage their emotions. Indeed, research shows that emotions contribute to an individual's ability to adapt to his environment by guiding him in social interactions (Keltner & Kring, 1998), by facilitating the detection of danger (Ohman et al., 2001), by preparing him to face a series of situations (Frijda, 1986), by accelerating and orienting his decision making (Bechara & Damasio, 2005) and by allowing him to memorize important elements more easily (Luminet & Curci, 2008). In this sense, the individual's skills in emotional regulation seem to be essential to his well-being.